CLINICAL TRIAL: NCT04315155
Title: Ph I Study to Evaluate the Safety and Efficacy of Belinostat in Combination With Nivolumab Alone and With Ipilimumab in Patients With Previously Treated Metastatic or Advanced Carcinomas Enriched for ARID1A Loss of Function (Lof) Mutation
Brief Title: Evaluating Safety & Efficacy Belinostat Combo w Nivo Alone & w Ipi in Patients w Treated Metastatic/Advanced Carcinomas w ARID1A Lof Mutation
Acronym: BENEFIT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study abandoned for funding issues
Sponsor: University of Utah (Other)
Collaborators: Bristol-Myers Squibb (Industry); Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI130490
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Metastatic Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma | interventions — belinostat; Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: This is an open-label Phase I trial designed to determine the phase 2 recommended dose (RP2D) of belinostat in combination with nivolumab with or without ipilimumab. Overall, the trial will assess dosing and safety of two regimens in the study population:
  * The double regimen: belinostat in combination with nivolumab;
  * The triplet regimen: belinostat in combination with nivolumab and ipilimumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Double Regimen (Experimental): belinostat in combination with nivolumab
  Interventions: Drug: Belinostat; Drug: nivolumab
- Triplet Regimen (Experimental): belinostat in combination with nivolumab and ipilimumab
  Interventions: Drug: ipilimumab; Drug: nivolumab; Drug: Belinostat

INTERVENTIONS:
Drug: Belinostat — Doublet Regimen Dose levels for Part 1:
  Belinostat Dose Level 1 (starting dose) 500 mg/m2 Dose Level 2 750 mg/m2 Dose Level 3 1000 mg/m2
  Arms: Double Regimen
Drug: nivolumab — Doublet Regimen Dose levels for Part 1 Nivolumab Dose Level 1 (starting dose) 360 mg Dose Level 2 360 mg Dose Level 3 360 mg
  Arms: Double Regimen
Drug: ipilimumab — Triplet and Doublet Regimen Dose Levels for Phase 2 Ipilimumab Doublet Dose n/a Triplet Dose 1 mg/kg
  Arms: Triplet Regimen
Drug: nivolumab — Triplet and Doublet Regimen Dose Levels for Phase 2 Nivolumab Doublet Dose 360 mg IV Triplet Dose 3 mg/kg
  Arms: Triplet Regimen
Drug: Belinostat — Triplet and Doublet Regimen Dose Levels for Phase 2 Belinostat Doublet Dose RP2D Triplet Dose RP2D
  Arms: Triplet Regimen

SUMMARY:
This is an open-label Phase I trial designed to determine the phase 2 recommended dose (RP2D) of belinostat in combination with nivolumab with or without ipilimumab.

DETAILED DESCRIPTION:
Overall, the trial will assess dosing and safety of two regimens in the study population:

* The double regimen: belinostat in combination with nivolumab;
* The triplet regimen: belinostat in combination with nivolumab and ipilimumab. The trial will consist of two parts: Part 1 will establish the RP2D of belinostat in combination with nivolumab (doublet regimen) and Part 2 will assess the safety of the RP2D of belinostat in combination with nivolumab (doublet regimen) and ipilimumab (triplet regimen). In Part 1, the recommended phase 2 dose of belinostat will be determined by using an single-patient accelerated titration design confirmed by a modified 3+3 design.

Once the RP2D of belinostat is confirmed in Part 1, Part 2 will open to the expansion of the doublet regimen and begin assessing the triplet regimen. The assessment of safety for the triplicate regimen will follow a Bayesian approach as described in the Statistical Analysis section and Appendix 2.

Due to the expected contrast in toxicity profiles between immediate toxicity from belinostat at various dose levels and immune mediated toxicity from the doublet and the triplet regimens, the definition of dose-limiting toxicities and the DLT evaluation periods will differ for each regimen (doublet vs. triplicate). Patients will be managed according to the regimen administered.

Statistical Hypotheses: Belinostat in combination with nivolumab alone and with ipilimumab is safe and effective in patients with previously treated metastatic or advanced carcinomas with or without ARID1A loss of function (lof) mutations.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Histologically confirmed solid tumor with metastatic disease or with unresectable, locally advanced disease
* Patients must have progressed on at least one prior therapy; and

  * Have no further standard of care options or the available options are associated with minimal overall survival benefit; or
  * Have no further clinically acceptable therapy; or
  * The patient has declined standard therapy.

The discussion regarding the choice of standard therapy offered, if available, and patient's choice and reason(s) to decline standard therapy should be documented clearly in the research chart.

Patients may have progressed on immune checkpoint inhibitor therapy.

* Part 1 and Part 2, Cohorts 1 and 2: Malignancy harboring ARID1A loss of function (lof) mutations as determined by the standard of care next-generation sequencing. The advanced solid tumors enrolled are anticipated to be, but not restricted to, urothelial carcinoma, gastrointestinal malignancies (gastric, colorectal, pancreatic), and gynecological malignancies (ovarian and endometrial).
* Part 2, Cohort 3: Malignancy without ARID1A loss of function (lof) mutation (ARID1A wild type).
* Subject must have measurable disease by RECIST 1.1 criteria by CT or MRI.
* ECOG Performance Status ≤ 2.
* Adequate organ function as defined as:

  * Hematologic:

    * Absolute neutrophil count (ANC) ≥ 1500/mm3
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 10 g/dL
  * Hepatic:

    * Total Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
    * AST(SGOT)/ALT(SGPT) ≤ 3 × institutional ULN
    * Patients with liver metastases will be allowed to enroll with AST and ALT levels ≤ 5 x ULN.
  * Renal:

    * Estimated creatinine clearance ≥ 30 mL/min by Cockcroft-Gault formula:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Highly effective contraception for both male and female subjects throughout the study and at least 4 months after last study treatment administration.
* Recovery to baseline or ≤ Grade 1 CTCAE v5.0 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Homozygous for UGT1A1*28 allele or Gilbert syndrome.
* Subject has received systemic antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any investigational therapy ≤ 14 days or within 5 half-lives before starting study treatment, whichever is shorter.
* Subject has received radiotherapy ≤ 14 days before the first dose of study treatment. Localized radiation therapy for the treatment of symptomatic bone metastasis is allowed during that timeframe.
* Subjects who have undergone major surgery ≤ 3 weeks before starting study drug or who have not fully recovered from major surgery.
* Diagnosis of any other malignancy within 2 years before study enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, and low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation, or castration) or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms is allowed.
* Known brain metastases or cranial epidural disease.

  --Note: Brain metastases or cranial epidural disease adequately treated with radiotherapy and/or surgery and stable for at least 4 weeks before the first dose of study treatment will be allowed on trial. Subjects must be neurologically asymptomatic and without corticosteroid treatment at the time of the first dose of study treatment.
* Current evidence of uncontrolled, clinically significant intercurrent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Congestive heart failure New York Heart Association Class 3 or 4, unstable angina pectoris, serious cardiac arrhythmias.
    * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic events, or thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) within 3 months before the first dose.
    * Uncontrolled hypertension defined as a sustained systolic blood pressure ≥ 160mmHg or a diastolic blood pressure ≥ 100mmHg despite optimal management.
    * Note: Patients with uncontrolled hypertension who are not optimally managed may be rescreened once controlled hypertension is achieved.
    * Patients with uncorrectable prolonged QTc (Bezet formula) > 480 msec or concomitant use of medications(s) with a known risk of inducing Torsade de Pointes if such treatment cannot be discontinued or switched to a different medication before starting the study drug.
    * Note: If a single ECG shows a QTc with an absolute value > 480 msec, two additional ECGs approximately 2 minutes apart must be performed within 30 minutes of the initial ECG, and the average of these three consecutive results for QTc will be used.
  * Adrenal insufficiency
* Subjects with congenital long QT syndrome.
* Patients currently on or who will require valproic acid for any medical condition during the study
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [except for diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the principal investigator
  * Patients with celiac disease controlled by diet alone
* Current or prior use of immunosuppressive medication within 14 days of cycle one day one, EXCEPT for the following permitted steroids:

  * Intranasal, inhaled, topical steroids, eye drops or local steroid injection (eg,intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography (CT) scan premedication).
* History of active primary immunodeficiency
* Known HIV infection with a detectable viral load at the time of screening.

  --Note: Patients on effective antiretroviral therapy with an undetectable viral load at the time of screening are eligible for this trial.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination, and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), or hepatitis C.

  --Note: Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Live attenuated vaccinations within 4 weeks of cycle one day one and while on trial is prohibited.
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.5.2. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur before the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
rate of dose limiting toxicities (DLTs) during defined DLT period | 9-12 months
  assess the recommended phase 2 dose of belinostat in combination with nivolumab in patients with advanced solid tumors harboring ARID1A mutations.
rate of intolerable refractory immune mediated adverse events assessed during the defined DLT evaluation period | 12-18 months
  assess the safety and tolerability of belinostat in combination with nivolumab with and without ipilimumab in patients with advanced solid tumors.

SECONDARY OUTCOMES:
frequency and characterization of Adverse Events (AE) | up to 5 years
  assess the safety of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors
• The rate of clinical benefit defined as the proportion of evaluable patients achieving stable disease, a partial response, or a complete response per RECIST 1.1 criteria | up to 5 years
  assess the efficacy of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors
• Objective response rate (ORR) as defined as the proportion of evaluable patients achieving a partial response or a complete response per RECIST 1.1 criteria. | up to 5 years
  assess the efficacy of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors
• Duration of response (DoR) as defined as the time from documented tumor response to disease progression as defined by RECIST 1.1. | up to 5 years
  assess the efficacy of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors
• Progression-free survival (PFS) as defined as the time from the initiation of study therapy to disease progression per RECIST 1.1, initiation of alternative therapy, or death from any cause. | up to 5 years
  assess the efficacy of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors
Overall survival (OS) | up to 5 years
  assess the efficacy of belinostat in combination with nivolumab with or without ipilimumab in patients with advanced solid tumors

IPD SHARING:
Plan to Share IPD: No